CLINICAL TRIAL: NCT06567522
Title: Comparative Assessment of Effectiveness and Safety of Lumbar Erector Spinae Plane Block (L-ESPB) Versus Absence of Locoregional Block in Hip Surgery
Brief Title: Comparative Assessment of Effectiveness and Safety of L-ESPB Versus Absence of Locoregional Block in Hip Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Álvaro Cunqueiro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ESPL - MORFINA
Record Dates: First submitted 2024-08-10; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Hip Fractures; Lumbar Erector Spinae Plane Block
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Pragmatic single-centre parallel group randomized clinical trial
Who Masked: Care Provider
Masking Description: Pragmatic randomized low interventional single-centre parallel non blinded design with blinded assessment of the objectives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ESP-L (Experimental): After hip fracture surgery ultrasound-guided ESP-L shall be carried out at the L3-14 level with 30 mL of levobupivacaine 0.25%
  Interventions: Drug: Lumbar Erector Spinae Plane Block. L bupivacaína 0.25%
- No ESP-L (No Intervention): Conventional intravenous analgesia after hip fracture surgery

INTERVENTIONS:
Drug: Lumbar Erector Spinae Plane Block. L bupivacaína 0.25% — Ultrasound-guided ESP-L shall be carried out at the L3-14 level with 30 mL of levobupivacaine 0.25%
  Arms: ESP-L

SUMMARY:
Hip surgery accounts for a high percentage of both emergency and elective surgical procedures in hospitals. Regardless of surgery being prescribed to treat a fracture or coxarthrosis, patients are usually elderly with multiple associated comorbidities. When faced with this patient profile, there is a tendency to undertreat pain for fear of the side effects and pharmacological interactions of conventional analgesic drugs.

Ultrasound-guided regional anesthesia applied in orthopedic and trauma surgery has been shown to reduce the doses of opioids and conventional analgesics, to ease deambulation and early recovery, to improve respiratory dynamics and to reduce vein thrombosis and pneumonias. Our study aims to verify whether L-ESP block is effective in the hip and proximal femur surgeries and allows to lower the dosage of opioids in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes over 18 years of age having undergone hip surgery
* ASA I-III (classification system used by the American Society of Anesthesiologists where I is low anesthetic risk and IV is high risk)
* Capacity to comprehend the principles of pain assessment using the VAS visual analogue scale
* Previously signed an informed consent.

Exclusion Criteria:

* Contraindications for the technique and/or the drugs used in this context
* Technical inability to perform the block
* Severe cognitive impairment or prior mental disabilities described in their medical records
* Patients already included in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-06-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the analgesic effectiveness and safety of lumbar ESP block versus absence of block after hip and proximal femur surgeries by means of the VAS scale with pain reduction of at least 1 point in the first two hours after surgery. | 2 hours after surgery
  Collect data on post-surgery pain using the Visual Analogue Scale (VAS).The VAS scale ranges from 0 to 10, with 0 being no pain and 10 being maximum pain.

SECONDARY OUTCOMES:
Compare the analgesic postoperative needs after performing L-ESP block versus a control group of patients having undergone hip or proximal femur surgeries and the postoperative consumption of opioids in both groups | 12 hours postoperative
  Consumption of morphine (mg)
Percentage of patients with technical ease to perform the esp-l block | 48 hours postoperative
  We will define the technical ease of the esp-l block from 1 to 3. 1 being good and when we are able to clearly distinguish anatomical structures in order to carry out the locoregional analgesia, 2 would be equivalent to regular, when these are sensed but not clearly defined structures and bad when we are not able to distinguish any anatomical structure that allows us to carry out the block.
Patient satisfaction survey on pain management | 48 hours postoperative
  We will classify patients into two groups according to their satisfaction with pain management in the postoperative period of hip surgery.
  Being the group of patients who consider themselves satisfied with pain management when it meets their expectations and dissatisfied if the patients are discomforted with it.
Describe de side effects of the lumbar ESP block and morphine | 48 hours postoperative
  pruritus, nausea, vomiting, erythema, hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Laura García Reza, Principal Investigator — Hospital Álvaro Cunqueiro
Locations (1):
- Hospital Álvaro Cunqueiro, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Garcia-Reza L, Raposeiras S, P Loureiro J, Pita-Romero R, Amate Pena JJ, Pereira Loureiro MA. Effectiveness and Safety of Lumbar Erector Spinae Plane Block Versus No Locoregional Block in Hip Surgery: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 15;14:e75854. doi: 10.2196/75854. PMID 40953436

DOCUMENTS (2):
  • Study Protocol (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT06567522/Prot_000.pdf
  • Informed Consent Form (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT06567522/ICF_001.pdf